CLINICAL TRIAL: NCT03785145
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Lateral Canthal Lines
Brief Title: MT10109L in the Treatment of Lateral Canthal Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT10109L-002; 2014-005279-10 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Lateral Canthal Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT10109L (Experimental): MT10109L will be injected into the LCL: initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period.
  Interventions: Drug: MT10109L
- Placebo (Placebo Comparator): Placebo will be injected into the LCL: initial double-blind treatment on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT10109L — MT10109L will be injected into the LCL.
  Other Names: NivobotulinumtoxinA
  Arms: MT10109L
Drug: Placebo — Placebo will be injected into the LCL.
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of MT10109L in the treatment of lateral canthal lines (LCL) in participants with moderate to severe LCL.

ELIGIBILITY:
Inclusion Criteria

• Female participants must not be pregnant or planning to get pregnant and willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.

Exclusion Criteria

* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of facial nerve palsy.
* Any uncontrolled systemic disease.
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study intervention).
* Anticipated need for surgery or overnight hospitalization during the study.
* Prior exposure to botulinum toxin of any serotype for any reason.
* Prior periorbital surgery, facial lift (full face or mid-face), thread lift, brow lift, or related procedures (eg, eyelid [blepharoplasty] and/or eyebrow surgery).
* Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol-specified study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMi Park, Study Director — Medytox Inc.
Locations (14):
- United States (9):
  - Advanced Research Associates, Glendale, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Skin Research Institute LLC, Coral Gables, Florida
  - Coleman Dermatologic Surgery Center, Metairie, Louisiana
  - MD Laser, Skin, & Vein Institute, Hunt Valley, Maryland
  - Laser Skin Surgery Center of New York, New York, New York
  - Bellaire Dermatology Associates, Bellaire, Texas
  - SkinDC, Arlington, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Russia (2):
  - Moscow scientific-practical centre of dermatovenerology and cosmetology, Moscow
  - State Budget Institution of Higher Education North-Western State Medical University named after I.I Mechnikov, Saint Petersburg
- United Kingdom (3):
  - Expert Aesthetics Ltd, Alderley Edge, Cheshire
  - Waverley Medical Practice, Coatbridge, North Lanarkshire
  - Medizen Clinic, Sutton Coldfield, West Midlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 235 met the inclusion/exclusion criteria and were randomized. 234 participants entered the study and were treated.
  This note is to explain why the number of participants to start a Period is not equal to the number who completed previous Period: Only participants who met the retreatment criteria received additional treatments (up to 2 times) in open label period. Therefore, the total number of treatments was different for each participant.
Groups:
- Placebo During Double-blind/MT10109L During Open-label: Placebo was injected into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1.
  Double-blind portion: Placebo was injected into the LCL.
  Open-label portion: In the open-label part, participants who met retreatment criteria were allowed up to 2 MT10109L injections
- MT10109L During Double-blind/MT10109L During Open-label: MT10109L was injected into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period.
  Double-blind portion: MT10109L was injected into the LCL. Open-label portion: Participants who met retreatment criteria were allowed up to 2 additional MT10109L injections
Period: Cycle 1 - Double Blind (Days 1-180)
Arm/Group | Placebo During Double-blind/MT10109L During Open-label | MT10109L During Double-blind/MT10109L During Open-label
Started | 77 (Note: 1 participant was randomized to the placebo group but was not treated. While 77 participants were randomized only 76 were treated in the placebo group.) | 158
Completed | 68 | 145
Not Completed | 9 | 13
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 1
Not completed — 1 participant was randomized to the placebo group but was not treated. This is counted in 'Other '. | 1 | 0
Period: Cycle 2 - Open Label Treatment 1
Arm/Group | Placebo During Double-blind/MT10109L During Open-label | MT10109L During Double-blind/MT10109L During Open-label
Started | 65 | 144
Completed | 61 | 130
Not Completed | 4 | 14
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 1 | 6
Not completed — COVID-19; Enrolled in a different study | 2 | 3
Period: Cycle 3 - Open Label Treatment 2
Arm/Group | Placebo During Double-blind/MT10109L During Open-label | MT10109L During Double-blind/MT10109L During Open-label
Started | 49 | 91
Completed | 49 | 88
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — COVID-19, Enrolled in a different study | 0 | 1

BASELINE CHARACTERISTICS:
Population: 235 participants were included in the Intent To Treat (ITT) population (77 participants in the placebo group and 158 participants in theMT10109L group).
Groups:
- Placebo: Placebo was injected into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1.
  Placebo: Placebo was injected into the LCL.
  In the open-label part, participants who met retreatment criteria were allowed up to 2 MT10109L
- MT10109L: MT10109L was injected into the Lateral Canthal Lines (LCL): initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period.
  MT10109L: MT10109L was injected into the LCL.
- Total: Total of all reporting groups
Arm/Group | Placebo | MT10109L | Total
Number analyzed (Participants) | 77 | 158 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 149 | 224
  >=65 years | 2 | 9 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (11.09) | 46.6 (11.43) | 46.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 127 | 188
  Male | 16 | 31 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 33 | 43
  Not Hispanic or Latino | 67 | 125 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 7 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 74 | 145 | 219
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS) According to INVESTIGATOR AND PARTICIPANT Assessments of Lateral Canthal Lines (LCL) Severity at Maximum Smile at Day 30
Description: The primary efficacy measure is a composite endpoint and a participant is considered responder only if both the investigator and participant independently report a ≥ 2-grade improvement at Day 30 of Double-Blind Period from baseline. Both participant and investigator used FWS to assess GL severity. FWS is 4-grade scale (0 to 3): 0=none, 1=mild, 2=moderate and 3=severe
Time Frame: Day 30
Population: All primary and secondary efficacy analyses endpoints were carried out using the Intent-To-Treat (ITT) analysis set, which was defined as all participants who were randomized. Multiple imputation method was used for missing variables in primary efficacy endpoint. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 77 | 158
Participants | 2 | 48

2. Secondary Outcome: The Percentage of Responders for INVESTIGATOR Assessments of Lateral Canthal Lines (LCL) Severity at Maximum Smile Using the Facial Wrinkle Scale (FWS)
Description: The Percentage of Responders for Investigator Assessments of Lateral Canthal Lines (LCL) Severity at Maximum Smile Using the Facial Wrinkle Scale (FWS), where a Responder was defined as Achieving a≥2-grade Improvement from Baseline at Maximum Smile at Day 30.
  The investigator evaluates the participant's LCL severity using a 4-point scale (0 to 3) where 0=none, 1=mild, 2=moderate and 3=severe.
Time Frame: Day 30
Population: All secondary efficacy analyses endpoints were carried out using the Intent-To-Treat (ITT) analysis subset at day 30, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 72 | 147
Participants | 3 | 57

3. Secondary Outcome: The Duration of Lateral Canthal Lines (LCL) Treatment in Participants Who Achieved a Rating of ≥ 2 Grade Improvement From Baseline in LCL Severity at Maximum Smile at Day 30 According to Investigator Assessments Using the Facial Wrinkle Scale (FWS)
Description: The investigator evaluates the participant's LCL severity using a 4-grade scale (0 to 3) where 0=none, 1=mild, 2=moderate and 3 = severe using the Facial Wrinkle Scale (FWS). The outcome is measured as median time to loss of treatment effect (i.e., return to moderate or severe LCL severity at maximum smile using the FWS).
Time Frame: Day 1 (first treatment) to Day 180
Population: The analysis population for this outcome includes the participants who achieved a rating of ≥ 2-grade improvement from baseline in LCL severity at maximum smile at Day 30 according to investigator assessments using the Facial Wrinkle Scale (FWS). This corresponds to the responders for Outcome 2. Note: Analyses of the secondary efficacy variables were performed using observed data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 3 | 57
Days | 242 [NA to NA] — The median duration and its 95% CI for placebo group was not meaningful as there were only 3 responders and therefore insufficient number of participants with events. | 148 [114.0 to 158]

4. Secondary Outcome: The Percentage of Participants Reporting Mostly Satisfied/Very Satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 for Lateral Canthal Lines (LCL)
Description: The Satisfaction Question 5 grades facial line treatment satisfaction on a 5-point scale (-2 to 2) where -2=Very dissatisfied and 2=Very satisfied.
Time Frame: Day 60
Population: All secondary efficacy analyses endpoints were carried out using the Intent-To-Treat (ITT) analysis subset at day 60, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 67 | 137
Participants | 4 | 107

5. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Lateral Canthal Lines (LCL) Severity at Rest Using the Facial Wrinkle Scale (FWS)
Description: The investigator evaluates the participant's LCL severity using a 4-point scale (0 to 3) where 0=none, 1=mild, 2=moderate and 3=severe.
  The outcome was measured among participants who were at least mild at rest at baseline, where a responder was defined as achieving a >=1-grade improvement from baseline at Day 30.
Time Frame: Day 30
Population: This secondary efficacy analysis was carried out using the Intent-To-Treat (ITT) analysis subset at day 30, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 71 | 135
Participants | 11 | 75

6. Secondary Outcome: Number of Patients Who Experienced an Adverse Event (AE) Through the Study Duration
Description: This section focuses primarily on Treatment Emergent Adverse Events(TEAEs), i.e., AEs that started or worsened after the first dose of study intervention (Day 1) until up to 30 days after their last visit or study exit. TEAE's are recorded by the PI and their study team from observations made after treatment administration. The safety analyses were conducted in the Safety population. Unless otherwise noted, safety results refer to TEAEs. All safety analyses were performed with participants analyzed by their actual treatment or regimen received.
Time Frame: AEs that started or worsen after the first dose of study intervention and up to 30 days after their last visit or study exit (Day 360 or early exit)
Population: All safety analyses were carried out using the Safety population set defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received.
  Please note: Participants in placebo group who entered open-label phase (post Day 180) and received study intervention (MT10109L) are counted in MT10109L group. Thus, overall number of participants in MT10109L group is greater than what is noted in participants flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 76 | 223
Participants | 12 | 78

7. Secondary Outcome: Mean Change From Baseline in Systolic Blood Pressure (BP)
Description: The outcome reported here is the mean change in Systolic BP from baseline to study exit.
Time Frame: Baseline to Day 360
Population: All safety analyses were carried out using the Safety population subset at study exit, defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received.
  In order to calculate the mean change from baseline, participants with non-missing analysis values at both baseline and post-baseline during that analysis visit were used.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 134
mmHg | 1.8 (12.28) | 0.5 (11.83)

8. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (BP)
Description: The outcome reported here is the mean change in Diastolic BP from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 134
mmHg | 0.4 (9.73) | 0.3 (9.42)

9. Secondary Outcome: Mean Change From Baseline in Pulse Rate
Description: The outcome reported here is the mean change in Pulse Rate from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 134
beats/min | -2.0 (13.13) | -0.8 (11.38)

10. Secondary Outcome: Mean Change From Baseline in Respiratory Rate
Description: The outcome reported here is the mean change in Respiratory Rate from baseline to study exit.
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 134
breaths/min | 0.7 (2.34) | -0.1 (1.89)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - Heart Rate
Description: The outcome reported here is a mean change in mean heart rate from baseline to studyexit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
beats/min | 2.9 (10.15) | 4.9 (10.36)

12. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - PR Interval
Description: The outcome reported here is a mean change in PR Interval from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | -2.1 (12.76) | -0.7 (13.65)

13. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QRS Duration
Description: The outcome reported here is a mean change in QRS duration from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | 2.6 (9.17) | 0.8 (7.14)

14. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QT Interval
Description: The outcome reported here is a mean change in QT Interval from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | -3.9 (22.08) | -11.3 (23.92)

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcB Interval
Description: The outcome reported here is a mean change in QTcB Interval from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | 3.7 (18.42) | 1.8 (20.3)

16. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcF Interval
Description: The outcome reported here is a mean change in QTcF Interval from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | 1.0 (14.97) | -2.9 (16.79)

17. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - RR Interval
Description: The outcome reported here is a mean change in RR Interval from baseline to study exit
Time Frame: Baseline to Day 360
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 66 | 126
milliseconds | -32.2 (122.66) | -58.2 (127.37)

18. Secondary Outcome: Number of Participants With Binding and Neutralizing Antibodies
Description: Only samples that tested positive in the binding antibody confirmatory assay were evaluated for neutralizing antibodies. The participants with positive neutralizing antibodies are only shown.
Time Frame: Baseline to Day 360
Population: The immunogenicity was analyzed in Safety population, defined as participants who received at least 1 dose of study intervention. Participants were grouped based on their actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 76 | 158
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: The time frame for the treatment-emergent adverse events(TEAEs) was from the first dose on Day 1 and up to 30 days after their last visit or study exit (Day 360 or early exit)
Description: All safety analyses were carried out using the Safety population, defined as participants who received at least 1dose of study intervention. Participants were grouped based on their actual treatment received and not planned treatment. TEAE's experienced by the participants in the placebo group during the open-label part (MT10109L Cycles 2 and 3) were counted in MT10109L group.
Arm/Group | Placebo | MT10109L
All-Cause Mortality (participants affected / at risk) | 0/76 | 1/223
Serious Adverse Events (participants affected / at risk) | 0/76 | 7/223
Other Adverse Events (participants affected / at risk) | 0/76 | 0/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | MT10109L (N=223)
Death (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General research agreement between the sponsor and PI's that includes a confidentiality section with a statement that the sponsor is and shall remain the exclusive owner of 'Information'. 'Information' shall include, but shall not be limited to, protocols, trade secrets, know-how, formulations, inventions, techniques, equipment, data and results.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT03785145/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03785145/SAP_001.pdf